CLINICAL TRIAL: NCT00237315
Title: Longitudinal Study of Urea Cycle Disorders
Status: Recruiting | Type: Observational
Sponsor: Andrea Gropman (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Rare Diseases Clinical Research Network (Network)
Responsible Party: Sponsor-Investigator, Andrea Gropman, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Other Study IDs: RDCRN 5101; U54RR019453 (NIH); U54HD061221 (NIH)
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Brain Diseases, Metabolic, Inborn; Amino Acid Metabolism, Inborn Errors; Urea Cycle Disorders
Keywords: Urea; Inherited metabolic disorders
MeSH Terms: conditions — Brain Diseases, Metabolic, Inborn; Amino Acid Metabolism, Inborn Errors; Urea Cycle Disorders, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants may elect to send a sample to the NIGMS Cell Repository at Coriell. Coriell establishes a cell line with the sample. These samples may be requested by investigators with a valid protocol. Requests should be directed to Coriell at nigms@coriell.org.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Urea cycle disorders (UCD) are a group of rare inherited metabolism disorders. Infants and children with UCD commonly experience episodes of vomiting, lethargy, and coma. The purpose of this study is to perform a long-term analysis of a large group of individuals with various UCDs. The study will focus on the natural history, disease progression, treatment, and outcome of individuals with UCD.

DETAILED DESCRIPTION:
Urea cycle disorders are a group of rare genetic diseases that affect how protein is broken down in the body. UCDs are caused by a deficiency in one of six enzymes or two mitochondrial membrane transporters responsible for removing ammonia, a waste product of protein metabolism, from the bloodstream. Normally, ammonia is converted into urea and then removed from the body in the form of urine. In UCDs, however, ammonia accumulates unchecked and is not removed from the body. It then reaches the brain through the blood, where it causes irreversible brain damage and/or death.

All UCDs, except for one (ornithine transcarbamylase deficiency), are inherited as recessive traits. The purpose of this study is to perform a long-term analysis of a large group of individuals with various UCDs. Biochemical status, growth, and cognitive function will be assessed. Survival and cognitive outcome of the two most commonly used forms of treatment, alternate pathway therapy and transplantation, will be evaluated. In addition, this study will identify the biochemical changes that may predict future metabolic imbalances so that they may be corrected before clinical symptoms develop.

This observational study is funded through 2025. All participants will attend an initial study visit, which will include a medical and diet history, physical and neurological examinations, psychological testing, and blood tests. Participants will then be followed with subsequent study visits, which will last 2-3 hours each. Individuals with neonatal onset UCD will be assessed every 3 months until age 2 and every 6 months thereafter. Individuals with late onset UCD will be evaluated every 6 months. Psychological testing will take place every 2 years. Psychological testing will take from 30 minutes (for younger children) up to 3 hours, depending on test battery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAGS deficiency, defined as the detection of a pathogenic mutation, and/or decreased (less than 20 % of control) NAGS enzyme activity in liver ,and/or hyperammonemia and first degree relative meets at least one of the criteria for NAGS deficiency
* Diagnosis of CPS I deficiency, defined as decreased (less than 20 % of control) CPS I enzyme activity in liver, and/or an identified pathogenic mutation, and/or hyperammonemia and first degree relative meets at least one of the criteria for CPS I deficiency
* Diagnosis of OTC deficiency, defined as the identification of a pathogenic mutation, and/or less than 20% of control of OTC activity in the liver, and/or elevated urinary orotate (greater than 20 uM/mM) in a random urine sample or after allopurinol challenge test, and/or hyperammonemia and first degree relative meets at least one of the criteria for OTC deficiency
* Diagnosis of AS deficiency (Citrullinemia), defined as a greater than or equal to 10-fold elevation of citrulline in plasma, and/or decreased AS enzyme activity in cultured skin fibroblasts or other appropriate tissue, and/or identification of a pathogenic mutation in the AS gene, and/or hyperammonemia and first degree relative meets at least one of the criteria for AS Deficiency
* Diagnosis of AL deficiency (Argininosuccinic Aciduria, ASA), defined as the presence of argininosuccinic acid in the blood or urine, and/or decreased AL enzyme activity in cultured skin fibroblasts or other appropriate tissue, and/or identification of a pathogenic mutation in the AL gene, and/or hyperammonemia and first degree relative meets at least one of the criteria for AL Deficiency
* Diagnosis of ARG deficiency (Hyperargininemia), defined as a greater than or equal to 5-fold elevated arginine levels in the blood, and/or decreased arginase enzyme levels in red blood cells or other appropriate tissue, and/or identification of a pathogenic mutation in the ARG gene, and/or hyperammonemia and first degree relative meets at least one of the criteria for ARG Deficiency
* Diagnosis of HHH Syndrome or ORNT deficiency, defined as a greater than or equal to 5-fold elevated plasma ornithine and homocitrulline levels in the urine, and/or a pathogenic mutation, and/or less than 20% residual labeled ornithine incorporation into protein in cultured fibroblasts, and/or hyperammonemia and first degree relative meets at least one of the criteria for HHH Syndrome or ORNT Deficiency
* Diagnosis of CITR deficiency (Citrullinemia Type II), defined as elevated citrulline levels in the blood and a pathogenic mutation and/or hyperammonemia and first degree relative meets criteria for CITR Deficiency
* Pending diagnosis of a UCD (UCD highly likely), defined as laboratory values highly suggestive of a UCD with symptomatic hyperammonemic episodes but without a verifiable diagnosis

Exclusion Criteria:

* Hyperammonemia caused by an organic academia, lysinuric protein intolerance, mitochondrial disorder, congenital lactic academia, fatty acid oxidation defects, or primary liver disease
* Rare and unrelated comorbidities (e.g., Down's syndrome, intraventricular hemorrhage in the newborn period, and extreme prematurity)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Enrollment goal: 1,100 participants
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2006-02 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of specific morbid indicators of disease severity | End of study
  hyperammonemia, developmental disabilities, long-term renal and hepatic effects, and case-fatality associated with the various forms of UCD
Relationship between various biomarkers and disease severity and progression | End of study
  correlation between glutamine, ammonia, liver function (biomarkers) and severity scale and IQ in terms of outcome
Safety and efficacy of currently used and new UCD therapies | End of study
  Interim events related to treatments (drugs, diet or liver transplant)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Gropman, MD, Study Chair — Children's National Research Institute; Susan Berry, MD, Study Chair — University of Minnesota Masonic Children's Hospital
Locations (15):
- United States (12):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Hospital Boston (UCDC New England Center), Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Case Western Medical College, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Children's Hospital and Regional Medical Center, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada
- University of Heidelberg, Heidelberg, Germany
- University Children's Hospital, Zurich, Switzerland

REFERENCES:
- [Background] Patrick TB, Richesson R, Andrews JE, Folk LC. SNOMED CT coding variation and grouping for "other findings" in a longitudinal study on urea cycle disorders. AMIA Annu Symp Proc. 2008 Nov 6;2008:11-5. PMID 18998949
- [Background] Richesson RL, Lee HS, Cuthbertson D, Lloyd J, Young K, Krischer JP. An automated communication system in a contact registry for persons with rare diseases: scalable tools for identifying and recruiting clinical research participants. Contemp Clin Trials. 2009 Jan;30(1):55-62. doi: 10.1016/j.cct.2008.09.002. Epub 2008 Sep 7. PMID 18804556
- [Background] Mitchell S, Ellingson C, Coyne T, Hall L, Neill M, Christian N, Higham C, Dobrowolski SF, Tuchman M, Summar M; Urea Cycle Disorder Consortium. Genetic variation in the urea cycle: a model resource for investigating key candidate genes for common diseases. Hum Mutat. 2009 Jan;30(1):56-60. doi: 10.1002/humu.20813. PMID 18666241
- [Background] Jain-Ghai S, Nagamani SC, Blaser S, Siriwardena K, Feigenbaum A. Arginase I deficiency: severe infantile presentation with hyperammonemia: more common than reported? Mol Genet Metab. 2011 Sep-Oct;104(1-2):107-11. doi: 10.1016/j.ymgme.2011.06.025. Epub 2011 Jul 13. PMID 21802329
- [Background] Wilson JM, Shchelochkov OA, Gallagher RC, Batshaw ML. Hepatocellular carcinoma in a research subject with ornithine transcarbamylase deficiency. Mol Genet Metab. 2012 Feb;105(2):263-5. doi: 10.1016/j.ymgme.2011.10.016. Epub 2011 Nov 7. PMID 22129577
- [Background] Burrage LC, Jain M, Gandolfo L, Lee BH; Members of the Urea Cycle Disorders Consortium; Nagamani SC. Sodium phenylbutyrate decreases plasma branched-chain amino acids in patients with urea cycle disorders. Mol Genet Metab. 2014 Sep-Oct;113(1-2):131-5. doi: 10.1016/j.ymgme.2014.06.005. Epub 2014 Jul 3. PMID 25042691
- [Background] Burrage LC, Sun Q, Elsea SH, Jiang MM, Nagamani SC, Frankel AE, Stone E, Alters SE, Johnson DE, Rowlinson SW, Georgiou G; Members of Urea Cycle Disorders Consortium; Lee BH. Human recombinant arginase enzyme reduces plasma arginine in mouse models of arginase deficiency. Hum Mol Genet. 2015 Nov 15;24(22):6417-27. doi: 10.1093/hmg/ddv352. Epub 2015 Sep 10. PMID 26358771
- [Background] Krivitzky LS, Walsh KS, Fisher EL, Berl MM. Executive functioning profiles from the BRIEF across pediatric medical disorders: Age and diagnosis factors. Child Neuropsychol. 2016;22(7):870-88. doi: 10.1080/09297049.2015.1054272. Epub 2015 Jul 6. PMID 26143938
- [Background] Waisbren SE, He J, McCarter R. Assessing Psychological Functioning in Metabolic Disorders: Validation of the Adaptive Behavior Assessment System, Second Edition (ABAS-II), and the Behavior Rating Inventory of Executive Function (BRIEF) for Identification of Individuals at Risk. JIMD Rep. 2015;21:35-43. doi: 10.1007/8904_2014_373. Epub 2015 Feb 25. PMID 25712381
- [Background] Kolker S, Dobbelaere D, Haberle J, Burgard P, Gleich F, Summar ML, Hannigan S, Parker S, Chakrapani A, Baumgartner MR; E-IMD Consortium. Networking Across Borders for Individuals with Organic Acidurias and Urea Cycle Disorders: The E-IMD Consortium. JIMD Rep. 2015;22:29-38. doi: 10.1007/8904_2015_408. Epub 2015 Feb 22. PMID 25701269
- [Background] Posset R, Garbade SF, Boy N, Burlina AB, Dionisi-Vici C, Dobbelaere D, Garcia-Cazorla A, de Lonlay P, Teles EL, Vara R, Mew NA, Batshaw ML, Baumgartner MR, McCandless SE, Seminara J, Summar M, Hoffmann GF, Kolker S, Burgard P; Additional individual contributors of the UCDC and the E-IMD consortium. Transatlantic combined and comparative data analysis of 1095 patients with urea cycle disorders-A successful strategy for clinical research of rare diseases. J Inherit Metab Dis. 2019 Jan;42(1):93-106. doi: 10.1002/jimd.12031. PMID 30740724
- [Background] Shapiro E, Bernstein J, Adams HR, Barbier AJ, Buracchio T, Como P, Delaney KA, Eichler F, Goldsmith JC, Hogan M, Kovacs S, Mink JW, Odenkirchen J, Parisi MA, Skrinar A, Waisbren SE, Mulberg AE. Neurocognitive clinical outcome assessments for inborn errors of metabolism and other rare conditions. Mol Genet Metab. 2016 Jun;118(2):65-9. doi: 10.1016/j.ymgme.2016.04.006. Epub 2016 Apr 14. PMID 27132782
- [Background] Summar ML, Koelker S, Freedenberg D, Le Mons C, Haberle J, Lee HS, Kirmse B; European Registry and Network for Intoxication Type Metabolic Diseases (E-IMD). Electronic address: http://www.e-imd.org/en/index.phtml; Members of the Urea Cycle Disorders Consortium (UCDC). Electronic address: http://rarediseasesnetwork.epi.usf.edu/ucdc/. The incidence of urea cycle disorders. Mol Genet Metab. 2013 Sep-Oct;110(1-2):179-80. doi: 10.1016/j.ymgme.2013.07.008. Epub 2013 Jul 18. PMID 23972786
- [Background] Waisbren SE, Cuthbertson D, Burgard P, Holbert A, McCarter R, Cederbaum S; Members of the Urea Cycle Disorders Consortium. Biochemical markers and neuropsychological functioning in distal urea cycle disorders. J Inherit Metab Dis. 2018 Jul;41(4):657-667. doi: 10.1007/s10545-017-0132-5. Epub 2018 Feb 8. PMID 29423830
- [Background] Waisbren SE, Stefanatos AK, Kok TMY, Ozturk-Hismi B. Neuropsychological attributes of urea cycle disorders: A systematic review of the literature. J Inherit Metab Dis. 2019 Nov;42(6):1176-1191. doi: 10.1002/jimd.12146. Epub 2019 Aug 1. PMID 31268178
- [Background] Lerner S, Anderzhanova E, Verbitsky S, Eilam R, Kuperman Y, Tsoory M, Kuznetsov Y, Brandis A, Mehlman T, Mazkereth R; UCDC Neuropsychologists; McCarter R, Segal M, Nagamani SCS, Chen A, Erez A. ASL Metabolically Regulates Tyrosine Hydroxylase in the Nucleus Locus Coeruleus. Cell Rep. 2019 Nov 19;29(8):2144-2153.e7. doi: 10.1016/j.celrep.2019.10.043. PMID 31747589
- [Background] Posset R, Gropman AL, Nagamani SCS, Burrage LC, Bedoyan JK, Wong D, Berry GT, Baumgartner MR, Yudkoff M, Zielonka M, Hoffmann GF, Burgard P, Schulze A, McCandless SE, Garcia-Cazorla A, Seminara J, Garbade SF, Kolker S; Urea Cycle Disorders Consortium and the European Registry and Network for Intoxication Type Metabolic Diseases Consortia Study Group. Impact of Diagnosis and Therapy on Cognitive Function in Urea Cycle Disorders. Ann Neurol. 2019 Jul;86(1):116-128. doi: 10.1002/ana.25492. Epub 2019 May 13. PMID 31018246
- [Background] Zielonka M, Kolker S, Gleich F, Stutzenberger N, Nagamani SCS, Gropman AL, Hoffmann GF, Garbade SF, Posset R; Urea Cycle Disorders Consortium (UCDC) and the European Registry and Network for Intoxication type Metabolic Diseases (E-IMD) Consortia Study Group. Early prediction of phenotypic severity in Citrullinemia Type 1. Ann Clin Transl Neurol. 2019 Sep;6(9):1858-1871. doi: 10.1002/acn3.50886. Epub 2019 Aug 30. PMID 31469252
- [Background] Burrage LC, Madan S, Li X, Ali S, Mohammad M, Stroup BM, Jiang MM, Cela R, Bertin T, Jin Z, Dai J, Guffey D, Finegold M; Members of the Urea Cycle Disorders Consortium (UCDC); Nagamani S, Minard CG, Marini J, Masand P, Schady D, Shneider BL, Leung DH, Bali D, Lee B. Chronic liver disease and impaired hepatic glycogen metabolism in argininosuccinate lyase deficiency. JCI Insight. 2020 Feb 27;5(4):e132342. doi: 10.1172/jci.insight.132342. PMID 31990680
- [Background] Zielonka M, Garbade SF, Gleich F, Okun JG, Nagamani SCS, Gropman AL, Hoffmann GF, Kolker S, Posset R; Urea Cycle Disorders Consortium (UCDC) and the European registry and network for Intoxication type Metabolic Diseases (E-IMD) Consortia Study Group. From genotype to phenotype: Early prediction of disease severity in argininosuccinic aciduria. Hum Mutat. 2020 May;41(5):946-960. doi: 10.1002/humu.23983. Epub 2020 Jan 30. PMID 31943503
- [Background] Nagamani SCS, Ali S, Izem R, Schady D, Masand P, Shneider BL, Leung DH, Burrage LC. Biomarkers for liver disease in urea cycle disorders. Mol Genet Metab. 2021 Jun;133(2):148-156. doi: 10.1016/j.ymgme.2021.04.001. Epub 2021 Apr 8. PMID 33846069
- [Background] Scharre S, Posset R, Garbade SF, Gleich F, Seidl MJ, Druck AC, Okun JG, Gropman AL, Nagamani SCS, Hoffmann GF, Kolker S, Zielonka M; Urea Cycle Disorders Consortium (UCDC) and the European registry and network for Intoxication type Metabolic Diseases (E-IMD) Consortia Study Group. Predicting the disease severity in male individuals with ornithine transcarbamylase deficiency. Ann Clin Transl Neurol. 2022 Nov;9(11):1715-1726. doi: 10.1002/acn3.51668. Epub 2022 Oct 10. PMID 36217298
- [Background] Sen K, Whitehead M, Castillo Pinto C, Caldovic L, Gropman A. Fifteen years of urea cycle disorders brain research: Looking back, looking forward. Anal Biochem. 2022 Jan 1;636:114343. doi: 10.1016/j.ab.2021.114343. Epub 2021 Oct 9. PMID 34637785
- [Background] Izem R, McCarter R. Randomized and non-randomized designs for causal inference with longitudinal data in rare disorders. Orphanet J Rare Dis. 2021 Nov 23;16(1):491. doi: 10.1186/s13023-021-02124-5. PMID 34814939
- [Background] Lerner S, Eilam R, Adler L, Baruteau J, Kreiser T, Tsoory M, Brandis A, Mehlman T, Ryten M, Botia JA, Ruiz SG, Garcia AC, Dionisi-Vici C, Ranucci G, Spada M, Mazkereth R, McCarter R, Izem R, Balmat TJ, Richesson R; Members of the UCDC; Gazit E, Nagamani SCS, Erez A. ASL expression in ALDH1A1+ neurons in the substantia nigra metabolically contributes to neurodegenerative phenotype. Hum Genet. 2021 Oct;140(10):1471-1485. doi: 10.1007/s00439-021-02345-5. Epub 2021 Aug 21. PMID 34417872
- [Background] McGowan M, Ferreira C, Whitehead M, Basu SK, Chang T, Gropman A. The Application of Neurodiagnostic Studies to Inform the Acute Management of a Newborn Presenting With Sarbamoyl Shosphate Synthetase 1 Deficiency. Child Neurol Open. 2021 Jan 22;8:2329048X20985179. doi: 10.1177/2329048X20985179. eCollection 2021 Jan-Dec. PMID 33644249
- [Background] Sen K, Castillo Pinto C, Gropman AL. Expanding Role of Proton Magnetic Resonance Spectroscopy: Timely Diagnosis and Treatment Initiation in Partial Ornithine Transcarbamylase Deficiency. J Pediatr Genet. 2021 Mar;10(1):77-80. doi: 10.1055/s-0040-1709670. Epub 2020 Apr 23. PMID 33552645
- [Background] Stergachis AB, Krier JB, Merugumala SK, Berry GT, Lin AP. Clinical utility of brain MRS imaging of patients with adult-onset non-cirrhotic hyperammonemia. Mol Genet Metab Rep. 2021 Mar 13;27:100742. doi: 10.1016/j.ymgmr.2021.100742. eCollection 2021 Jun. PMID 33763331
- [Background] Murali CN, Barber JR, McCarter R, Zhang A, Gallant N, Simpson K, Dorrani N, Wilkening GN, Hays RD, Lichter-Konecki U; Members of the Urea Cycle Disorders Consortium; Burrage LC, Nagamani SCS. Health-related quality of life in a systematically assessed cohort of children and adults with urea cycle disorders. Mol Genet Metab. 2023 Nov;140(3):107696. doi: 10.1016/j.ymgme.2023.107696. Epub 2023 Sep 8. PMID 37690181
- [Background] Posset R, Zielonka M, Gleich F, Garbade SF, Hoffmann GF, Kolker S; Urea Cycle Disorders Consortium (UCDC) and European registry and network for Intoxication type Metabolic Diseases (E-IMD) Consortia Study Group. The challenge of understanding and predicting phenotypic diversity in urea cycle disorders. J Inherit Metab Dis. 2023 Nov;46(6):1007-1016. doi: 10.1002/jimd.12678. Epub 2023 Oct 10. PMID 37702610
- [Result] Tuchman M, Lee B, Lichter-Konecki U, Summar ML, Yudkoff M, Cederbaum SD, Kerr DS, Diaz GA, Seashore MR, Lee HS, McCarter RJ, Krischer JP, Batshaw ML; Additional members of Urea Cycle Disorders Consortium of the Rare Diseases Clinical Research Network. Cross-sectional multicenter study of patients with urea cycle disorders in the United States. Mol Genet Metab. 2008 Aug;94(4):397-402. doi: 10.1016/j.ymgme.2008.05.004. Epub 2008 Jun 17. PMID 18562231
- [Result] Krivitzky L, Babikian T, Lee HS, Thomas NH, Burk-Paull KL, Batshaw ML. Intellectual, adaptive, and behavioral functioning in children with urea cycle disorders. Pediatr Res. 2009 Jul;66(1):96-101. doi: 10.1203/PDR.0b013e3181a27a16. PMID 19287347
- [Result] Morgan TM, Schlegel C, Edwards KM, Welch-Burke T, Zhu Y, Sparks R, Summar M; Urea Cycle Disorders Consortium. Vaccines are not associated with metabolic events in children with urea cycle disorders. Pediatrics. 2011 May;127(5):e1147-53. doi: 10.1542/peds.2010-1628. Epub 2011 Apr 11. PMID 21482610
- [Result] Ah Mew N, Krivitzky L, McCarter R, Batshaw M, Tuchman M; Urea Cycle Disorders Consortium of the Rare Diseases Clinical Research Network. Clinical outcomes of neonatal onset proximal versus distal urea cycle disorders do not differ. J Pediatr. 2013 Feb;162(2):324-9.e1. doi: 10.1016/j.jpeds.2012.06.065. Epub 2012 Aug 15. PMID 22901741
- [Result] Seminara J, Tuchman M, Krivitzky L, Krischer J, Lee HS, Lemons C, Baumgartner M, Cederbaum S, Diaz GA, Feigenbaum A, Gallagher RC, Harding CO, Kerr DS, Lanpher B, Lee B, Lichter-Konecki U, McCandless SE, Merritt JL, Oster-Granite ML, Seashore MR, Stricker T, Summar M, Waisbren S, Yudkoff M, Batshaw ML. Establishing a consortium for the study of rare diseases: The Urea Cycle Disorders Consortium. Mol Genet Metab. 2010;100 Suppl 1(Suppl 1):S97-105. doi: 10.1016/j.ymgme.2010.01.014. Epub 2010 Feb 10. PMID 20188616
- [Result] Gallagher RC, Lam C, Wong D, Cederbaum S, Sokol RJ. Significant hepatic involvement in patients with ornithine transcarbamylase deficiency. J Pediatr. 2014 Apr;164(4):720-725.e6. doi: 10.1016/j.jpeds.2013.12.024. Epub 2014 Jan 30. PMID 24485820
- [Result] Batshaw ML, Tuchman M, Summar M, Seminara J; Members of the Urea Cycle Disorders Consortium. A longitudinal study of urea cycle disorders. Mol Genet Metab. 2014 Sep-Oct;113(1-2):127-30. doi: 10.1016/j.ymgme.2014.08.001. Epub 2014 Aug 10. PMID 25135652
- [Result] McGuire PJ, Lee HS; members of the Urea Cycle Disorders Consoritum; Summar ML. Infectious precipitants of acute hyperammonemia are associated with indicators of increased morbidity in patients with urea cycle disorders. J Pediatr. 2013 Dec;163(6):1705-1710.e1. doi: 10.1016/j.jpeds.2013.08.029. Epub 2013 Sep 29. PMID 24084106
- [Result] Waisbren SE, Gropman AL; Members of the Urea Cycle Disorders Consortium (UCDC); Batshaw ML. Improving long term outcomes in urea cycle disorders-report from the Urea Cycle Disorders Consortium. J Inherit Metab Dis. 2016 Jul;39(4):573-84. doi: 10.1007/s10545-016-9942-0. Epub 2016 May 23. PMID 27215558
- See also: Urea Cycle Disorders Consortium website — https://www.rarediseasesnetwork.org/cms/UCDC